CLINICAL TRIAL: NCT05660551
Title: Effect of Different Training Techniques in Teaching the Management of Shoulder Dystocia
Brief Title: Investigation of the Effect of Different Training Techniques in Teaching the Management of Shoulder Dystocia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, İlknur Münevver Gönenç, Associate Professor Dr., Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 737219
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Shoulder Dystocia
MeSH Terms: conditions — Shoulder Dystocia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention)
- Demonstration group (Experimental)
  Interventions: Other: Demostration
- Telesimulation Group (Experimental)
  Interventions: Other: Telesimulation
- Kahoot Game Group (Experimental)
  Interventions: Other: Kahoot Game

INTERVENTIONS:
Other: Demostration — This group will be demonstrated on a model after the theoretical training. The maneuvers used in the management of shoulder dystocia will be shown to the students on the model, respectively.
  Arms: Demonstration group
Other: Telesimulation — After the theoretical training for this group, telesimulation will be applied. A scenario will be created for the telesimulation experience and a video will be shot with this scenario. These videos will be watched by the students in groups of 4 on Microsoft Teams and a case discussion will be made through this scenario.
  Arms: Telesimulation Group
Other: Kahoot Game — Kahoot, a game-based program, will be applied to this group one week after the theoretical training. The game will be organized according to the learning objectives and achievements related to shoulder dystocia.
  Arms: Kahoot Game Group

SUMMARY:
In this study, it was aimed to determine the effect of demonstration, telesimulation and game-based teaching on teaching shoulder dystocia management in midwifery students.

H01: There is no difference between the four groups in terms of satisfaction with learning.

H02: There is no difference between the four groups in terms of Self-Confidence in Learning.

H03: There is no difference between the four groups in terms of Motivation scores in Teaching Materials.

ELIGIBILITY:
Inclusion Criteria:

* Being a registered student in the midwifery department,
* Having the ability to manage normal birth,
* Having a smart phone, tablet or computer with internet connection,
* Agreeing to participate in the research

Exclusion Criteria:

* to suspend education.
* Having received formal training on shoulder dystocia management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Dystocia Skill Checklist | 15 days after the training
  The skill checklist prepared by the researcher by scanning the literature consists of three parts (Taşkın, 2016; Sayıner & Başkaya, 2020); diagnosing shoulder dystocia, making the necessary interventions for shoulder dystocia at birth, and intervention after birth.In the skill list, the student will receive 1 point for each correct application, and 0 points for each incorrect or skipped application.Higher scores indicate higher skill levels.
Instructional Materials Motivation Survey | 15 days after the training
  The Instructional Materials Motivation Survey (IMMS) aims to assess the motivational characteristics of instructional materials or courses using the Attention, Relevance, Confidence, and Satisfaction (ARCS) model of motivation. The five-point Likert type scale consists of 36 items in the original scale.
  In the last Turkish adaptation study, 3 of the items were excluded from the original scale and a total of 33 items were included in the Turkish version of the scale.
Change in Self-Sufficiency | immediately before the training, immediately after the training
  Visual Analog Scale (VAS)- assessed by adequate vision. For each item, students rated their sense of self-sufficiency on a scale of 0 (very inadequate) to 10 (very adequate).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided